CLINICAL TRIAL: NCT05365893
Title: Window of Opportunity for Neoadjuvant Stroma Modification in Pancreatic Cancer
Brief Title: PHL Treatment in Pancreatic Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-1085; GI-174 (Other: Fox Chase Cancer Center); 1R21CA252535-01A1 (NIH)
Record Dates: First submitted 2021-11-04; First posted 2022-05-09 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: chemo-resistant cancer
MeSH Terms: interventions — paricalcitol; Hydroxychloroquine; Losartan; Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: 20 patients diagnosed with resectable pancreatic cancer will be consented for blood and tissue prior to starting neoadjuvant therapy.
  10 patients will be assigned to the experimental (PHL) arm (Arm A).
  Treatment arm; N=10 (Consented for PHL the time of neoadjuvant therapy completion): Experimental therapy 4-8 weeks pre-op:
  Paricalcitol 25 mcg IV administered M-W-F Hydroxychloroquine 600 mg PO BID Losartan 50 mg PO daily
  Control arm (Arm B); N=10 These patients have already signed consent for blood and tissue- will proceed to surgery at completion of neoadjuvant therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PHL (Paricalcitol, Hydroxychloroquine, Losartan) (Experimental): Paricalcitol 25 mcg IV administered M-W-F Hydroxychloroquine 600 mg PO BID Losartan 50 mg PO daily
  Interventions: Combination Product: Paricalcitol, Hydroxychloroquine, Losartan
- Neoadjuvant therapy and surgery only (Control) (Active Comparator): Control arm These patients will proceed to surgery at completion of neoadjuvant therapy.
  Interventions: Other: Neoadjuvant therapy and surgery only (Control)

INTERVENTIONS:
Combination Product: Paricalcitol, Hydroxychloroquine, Losartan — Paricalcitol 25 mcg IV administered M-W-F Hydroxychloroquine 600 mg PO BID Losartan 50 mg PO daily
  Arms: PHL (Paricalcitol, Hydroxychloroquine, Losartan)
Other: Neoadjuvant therapy and surgery only (Control) — Control arm These patients will proceed to surgery at completion of neoadjuvant therapy.
  Arms: Neoadjuvant therapy and surgery only (Control)

SUMMARY:
This proposal will investigate the effect of paricalcitol, hydroxychloroquine, and losartan (PHL) combination of 3 stroma-modifying drugs on pancreatic adenocarcinoma and its stroma.

DETAILED DESCRIPTION:
This study will test the feasibility and safety of these pancreatic ductal adenocarcinoma (PDAC) stroma modulators in the pre-operative setting, and will offer the opportunity to detect the combined effect on PDAC tissue constituents to validate the mechanism using real-time biologic end points. The long-term goal for PHL is to deploy this regimen in combination with chemotherapy to treat PDAC. Further, this study will establish a paradigm of a "window" trial (the use of novel therapies in the period of time between the end of neoadjuvant treatment and surgery) to test new compounds and establish their biological activities in PDAC.

This pilot trial will establish the feasibility and determine the biological activity of PHL combination given prior to surgery to 10 patients who completed neoadjuvant therapy (NAT) with modified FOLFIRINOX and chemoradiation using sequential blood and tissue samples (blood samples will be collected pre NAT and post chemotherapy; post chemoradiation; pre-surgery and post-surgery) and compare with 10 patients who undergo the same neoadjuvant therapy (modified FOLFIRINOX followed by chemo-RT and proceed to surgery without treatment with PHL regimen (blood sample in this group will be collected pre NAT and post-chemotherapy; post-chemoradiation, pre-surgery and post-surgery).

This is a single site pilot study of PHL in patients with resectable non-metastatic PDAC.

Study will enroll 20 patients who will be consented prior to initiation of NAT to donate blood (pre NAT, post neoadjuvant chemotherapy and post neoadjuvant radiation and pre and post-surgery) and tissue (archival tissue from diagnosis biopsy and surgical specimen). All patients will complete a minimum of 3 months of modified FOLFIRINOX + chemoradiation. Of these 20 patients, 10 will receive the study PHL regimen (Arm A) and 10 will serve as the control arm (Arm B).

10 patients will be treated with resectable non-metastatic PDAC with a combination of three stroma-modifying agents PHL during the "window of opportunity", spanning 4-8 weeks after conclusion of neoadjuvant chemotherapy plus radiation and prior to surgery (Fig 1). Neoadjuvant chemotherapy will consist of at least 3 months of modified FOLFIRINOX regimen followed by chemoradiotherapy. The choice of chemotherapy given concurrently with radiation will be at the discretion of the medical team and the patient. Patients should start on the trial medications at least 4 weeks prior to surgery and continue to take the medication until the day before surgery. All the patients in the treatment arm must receive PHL for a minimum of 4 weeks and for a maximum period of 8 weeks. Patients who discontinue before completing 4 weeks of therapy due to disease progression may be replaced.

ELIGIBILITY:
Inclusion Criteria for all study participants:

* Patients must have new diagnosed histologically or cytologically confirmed pancreatic adenocarcinoma.
* Patients must have resectable non-metastatic PDAC and anticipate receiving surgery in a minimum of 4 weeks and a maximum of 12 weeks from completing neoadjuvant chemotherapy and radiation.
* Patients are planned for a minimum of 3 months of modified FOLFIRINOX treatment followed by chemo/radiation followed by surgical resection.
* Age > 18 years.
* ECOG performance status 0-1
* Patients must have normal organ function as defined below
* Total bilirubin within normal institutional limits
* AST/ALT (SGOT/SGPT) < 5 times institutional normal limits
* Creatinine within normal institutional limits OR
* Creatinine clearance > 30 Ml/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential must be non-pregnant (negative pregnancy test within 72 hours prior to registration). Postmenopausal woman must have been amenorrhoeic and nonlactating for at least 12 months to be considered of non-childbearing potential. Men and women of child bearing potential must be willing to exercise an effective form of birth control (abstinence/contraception) while on study and for 3 months after therapy is completed.
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria for all study participants:

* Tumors of acinar or adenocarcinoma histology
* Patients may not be receiving any other investigational agents
* Patients currently receiving hydroxychloroquine or an angiotensin II receptor blocker
* Patients with radiological or cytologically confirmed metastatic or unresectable disease
* Pregnant or breast feeding. Refer to section 4.4 for further detail.

Inclusion criteria for participation in experimental PHL therapy (Arm A):

* Patients must have resectable non-metastatic PDAC and anticipate receiving surgery in a minimum of 4 weeks and a maximum of 12 weeks from completing neoadjuvant chemotherapy and chemoradiation.
* Patients completed a minimum of 3 months of modified FOLFIRINOX treatment followed by chemoradiation prior to study enrollment and plans for surgical resection.
* Ability to understand and willingness to sign a written informed consent and HIPAA consent document

Exclusion Criteria for participation in Experimental PHL Therapy (Arm A):

* Patients who have residual grade 3 or higher adverse events from prior chemotherapy or chemoradiotherapy for pancreatic cancer
* Concomitant use of an ACE inhibitor or ARB, vitamin D, or hydroxychloroquine. Patient may elect to stop Vitamin D supplement and will be allowed to enroll on the study.
* Patients cannot have a history of retinopathy, macular degeneration or other severe ocular issues, baseline hypotension (systolic blood pressure lower than 100 mmHg on two separate readings obtained on two separate days), or history of hypercalcemia requiring treatment
* Patients with known disorders precluding use of any of the study drugs including a history of angioedema, hypotension, or renal disease (CrCl < 30mL/min).
* History of allergic reactions attributed to compound of similar chemical or biologic composition to the agent(s) used in this study
* Patients receiving any medications or substances that significantly interact with PHL are ineligible (specified in section 5.2).
* A marked baseline prolongation of QT/QTc interval
* A history of additional risk factors for Torsades de Pointes (e.g., heart failure, family history of Long QT Syndrome)
* Atrio-ventricular blockade of 2nd or 3rd degree
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experience grade 3 or greater treatment-related adverse events assessed by CTCAE v5.0 | 4 weeks
  Feasibility of administering PHL when given in the window between neoadjuvant chemo-radiotherapy and surgery. Feasibility is defined as the ability to tolerate a minimum of 4 weeks of PHL treatment without interfering with patient's planned surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Reddy, MD, FACS, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No